CLINICAL TRIAL: NCT04160923
Title: Incidence and Neonatal Outcome of Eclamptic Parturient : a 13-years Retrospective Study From a Single Tertiary Care Center Anesthetic Aspect.
Brief Title: Incidence and Neonatal Outcome of Eclamptic Parturient in Tertiary Hospital.
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Pattrapun Wongsripuemtet, Principal Investigator, Siriraj Hospital
Other Study IDs: SIRB 390/2017
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Eclampsia
MeSH Terms: conditions — Eclampsia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eclampsia is a rare but serious disease that can happen during the pregnancy. Both general and regional anesthesia can both be performed in eclamptic patients. Eclamptic patients has greater risk if undergo general anesthesia such as risks associated with general anesthesia in pregnancy and also cerebral hemorrhage risks from hypertension during laryngoscope application and thrombocytopenia that can happen in eclamptic patients. So, most of Anesthesiologists tend to avoid performing general anesthesia in these patients. But spinal anesthesia also has side effects such as hypotension or epidural hematoma. And nowadays there's minimal evidence on suitable anesthesia in eclamptic patients. Our study wants to review on how choice of anesthesia affects these patients both mothers and their neonates

ELIGIBILITY:
Inclusion Criteria:

* Patient who diagnosed with eclampsia.

Exclusion Criteria:

* Incomplete medical record.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient who diagnosed with eclampsia during January2005-December 2017
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
The incidence of eclampsia in Siriraj Hospital. | 13 years
  Incidence represent as percent.

CONTACTS AND LOCATIONS:
Overall Officials: Soawaphak Chumpathong, Assoc. Prof., Study Director — Department of Anesthesiology, Siriraj Hospital, Mahidol University
Locations (2):
- Thailand (2):
  - Department of Anesthesiology, Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok
  - Pattrapun Wongsripuemtet, Bangkok Noi, Bangkok